CLINICAL TRIAL: NCT02492139
Title: ESP II Evaluation of the Reliability and Usability of the Reusable "BrownieForSymphony" Pump Set in Home Use
Brief Title: Evaluation of the Reliability and Usability of the Reusable "BrownieForSymphony" Pump Set in Home Use
Acronym: ESPII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medela AG (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: MBF1503
Record Dates: First submitted 2015-07-01; First posted 2015-07-08 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Lactation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pumping (Other): Each particpant will pump with the current pumpset one week and then two weeks with the pumpset
  Interventions: Device: Pumping CE-marked Symphony Pumpset; Device: Pumping BrownieForSymphony Pumpset

INTERVENTIONS:
Device: Pumping CE-marked Symphony Pumpset — Pumping with the CE-marked Symphony Pumpset
Device: Pumping BrownieForSymphony Pumpset — Pumping with the the BrownieForSymphony Pumpset

SUMMARY:
The overall purpose of this study is to evaluate the reliability and usability of the reusable BrownieForSymphony pump set in home use.

The primary objectives of this study is to asses and compare the System Usability Scale (SUS) score of the BrownieForSymphony pump set and the current used Symphony pump set.

Secondary Objectives

The secondary objectives of this study are:

to evaluate the rate of usability problems with the BrownieForSymphony pump set

* to evaluate the pragmatic quality (task/goal fulfilment) of the BrownieForSymphony pump set
* to evaluate perceived comfort during pumping with the BrownieForSymphony pump set Prospective Cohort Study (quasi Cross over design)

ELIGIBILITY:
Inclusion Criteria:

* Lactating woman >18 years who

  * Have been pumping for at least 7 days with the Symphony pump and pump set prior to study participation
  * Have been pumping at least 10 times in the week prior to study participation
  * Consistently pump 10 ml of milk or more per breast, per pumping session prior to study participation
  * Currently use a breast shield size of 24 mm
  * Participant has agreed to pump at least 10 times a week over the next three weeks

Exclusion Criteria:

* o Woman has a medical condition of the breast (eg. Mastitis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Usability Scale (SUS) Symphony Pumpset usability | after 7 days
  Rating of the Usability of the Symphony Pumpset
Usability Scale (SUS) BrownieForSymphony Pumpset usability | after 14 days
  Rating of the Usability of the Symphony Pumpset

SECONDARY OUTCOMES:
User experience questionnaire (UEQ) | after 7 days, 14 days, 3 week

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Steinfelder, Principal Investigator — Medela AG
Locations (1):
- Medela AG, Baar, Canton of Zug, Switzerland